CLINICAL TRIAL: NCT03705078
Title: A Multicenter Randomized Clinical Trial Comparing Two Treatment Strategies to Prevent Rebleeding From Gastric Varices: "Early TIPS" Versus Glue Obliteration
Brief Title: "Early TIPS" Versus Glue Obliteration to Prevent Rebleeding From Gastric Varices
Acronym: GAVAPROSEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/2018/76
Record Dates: First submitted 2018-10-09; First posted 2018-10-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Bleeding Gastric Varices; Cirrhosis
Keywords: Bleeding gastric varices; cirrhosis; type 2 gastro-esophageal varices; isolated gastric varices; transjugular intra-hepatic porto systemic shunt (TIPS); portal hypertension; glue obliteration; tissue adhesive
MeSH Terms: conditions — Fibrosis; Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early TIPS (Other): Transjugular portosytemic shunt within 72h
  Interventions: Procedure: Transjugular Portosytemic Shunt (TIPS)
- Glue obliteration (Other): glue obliteration repeated sessions
  Interventions: Procedure: glue obliteration

INTERVENTIONS:
Procedure: Transjugular Portosytemic Shunt (TIPS) — The TIPS is placed under radiologic guidance. A branch of the intrahepatic portal vein is punctured; afterwards, the splenic vein is catheterized so that a portal venography and pressure measurements can be performed. Then, the parenchymal track is dilated and a stent is placed. A final portography and pressure measurement in the main portal vein and the inferior caval vein are performed.
  Arms: early TIPS
Procedure: glue obliteration — The standard protocol uses cyanoacrylate and lipiodol in 1:1 ratio injecting with no more than 1 mL at the varix each time. In most cases, cyanoacrylate is usually extruded into the stomach lumen within 1-3 months after injection. The French observational survey observed that a large majority (78%) of practitioners diluted glue with lipiodol and most (68%) proposed a proportion of glue to lipiodol of 1:1 the total volume injected per varix (from 1mL to 20 mL) varied substantially. Regarding the type of glue, although the majority of published data concern Histoacryl®, nearly half of practitioners used Glubran®. This lack of preference for one glue over the other may be explained by the fact that only Glubran® is approved in this indication in Europe.
  Arms: Glue obliteration

SUMMARY:
The primary objective of the study is to demonstrate the superiority of an "early tips" strategy over standard treatment by glue obliteration (G0) in preventing bleeding recurrence or death at one year after a non GOV1 gastric variceal bleeding in cirrhotic patients initially treated by GO.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients: the diagnosis of liver cirrhosis will be based on previous needle liver biopsy or on the combination of clinical, biochemical, and radiological findings. If biopsy findings are unavailable and in case of non-complicated cirrhosis, non-invasive markers will be used.
* Variceal bleeding at endoscopy from gastroesophageal gastric varices type 2 or isolated gastric varices type 1 or 2 (Sarin classification) according to the following criteria: endoscopic signs of an active spurting or oozing from gastric varices (GV); adherent blood clots, white nipple signs, or erosions on the GV and absence of other bleeding sources.
* Hemodynamically stable patient (Mean arterial pressure above 65 mmHg) without clinical significant rebleeding (Baveno criteria) within 12 hours after the initial endoscopy with glue obliteration.
* Written informed consent obtained.

Exclusion Criteria:

* Pregnant woman or breastfeeding.
* Minor and patients older than 75 years.
* Non cirrhotic portal hypertension.
* Hepatocellular carcinoma outside the Milan criteria or other cancer at a palliative stage.
* Child Pugh score > 13.
* History of severe or refractory hepatic encephalopathy unrelated to gastrointestinal bleeding.
* Congestive heart failure.
* History or presence of pulmonary hypertension.
* Patients with other indication for TIPS.
* Uncontrolled gastric variceal bleeding.
* Portal vein cavernoma.
* Patient who have previously received a TIPS procedure.
* Failure to receive clear information in patients without an identified trusted person.
* Refusal of the participation agreement by signing the information form and consent as defined.
* Exclusion period from another biomedical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant rebleeding (upper gastrointestinal bleeding whatever its origin) | 12 months
  Defined by Baveno VI consens group as a recurrent melena or hematemesis resulting in any of the following:
  * Hospital admission
  * Blood transfusion
  * 3 g/dL drop in hemoglobin
death | 12 months

SECONDARY OUTCOMES:
All-cause mortality and liver-related mortality | Day 42
All-cause mortality and liver-related mortality | 12 months
Incidence of rebleeding | Day 42
Incidence of rebleeding | Day 90
Incidence of rebleeding | 3 months
Incidence of rebleeding | 12 months
Cumulative number of packed red blood cells | Day 42
Cumulative number of packed red blood cells | 12 months
Incidence of complications of cirrhosis (infections, ascites, hepatic encephalopathy, hepatorenal syndrome) during follow-up | 12 months
Frequency of TIPS complications | 12 months
Frequency of glue obliteration complications | 12 months
MELD score (Model for End Stage Liver Disease) in TIPS group | 6 months
  MELD score = 9.57*LN(creatinin in mg/dl) + 3.78*LN(Bilirubin in mg/dl) + 11.2*LN(INR) + 6.43
MELD score (Model for End Stage Liver Disease) in glue obliteration group | 6 months
  MELD score = 9.57*LN(creatinin in mg/dl) + 3.78*LN(Bilirubin in mg/dl) + 11.2*LN(INR) + 6.43
Number of days of hospitalization | 12 months

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Besançon, Besançon
  - Univerity Hospital of Bondy, Bondy
  - University Hospital of Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - University Hospital of Caen, Caen
  - University Hospital of Dijon, Dijon
  - University Hospital of Lille, Lille
  - CHU Lyon, Lyon
  - University Hospital of Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - Pitié Salpétrière Hospital, Paris
  - St Antoine Hospital, Paris
  - University Hospital of Rennes, Rennes
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tours, Tours
  - Paul Brousse Hospital, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cervoni JP, Weil D, Desmarets M, Lannes A, D'Alteroche L, Bouzbib C, Larrue H, Lemaitre E, Faure S, Latournerie M, Jezequel C, Billioud C, Carbonell N, Saliba F, Tanne F, Hiriart JB, Olivier-Hourmand I, Nguyen Khac E, Archambeaud I, Hilleret MN, Oberti F, Elkrief L, Meunier L, Gerster T, Rode A, Bardou-Jacquet E, Robic MA, Ozenne V, Sacleux SC, Reboux N, Chermak F, Calame P, Borentain P, Thevenot T, Di Martino V, Thabut D, Louvet A, Rudler M, Bureau C; le Club Francophone pour l'Etude de l'Hypertension Portale, and the GAVAPROSEC study group. Pre-emptive TIPS for gastric variceal bleeding in patients with cirrhosis (GAVAPROSEC): an open-label randomised clinical trial. Lancet Gastroenterol Hepatol. 2025 Aug;10(8):726-733. doi: 10.1016/S2468-1253(25)00156-6. Epub 2025 Jun 12. PMID 40517780

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03705078/SAP_000.pdf